CLINICAL TRIAL: NCT00131898
Title: Phase III Prospective Randomized Trial of Pre-Operative Intensity Modulated Radiation Therapy (IMRT) Plus Surgery Versus Surgery Alone For Primary Retroperitoneal Sarcoma
Brief Title: A Prospective Randomized Trial of Pre-Operative IMRT+Surgery Versus Surgery Alone For Primary Retroperitoneal Sarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Samuel Singer, MD, Memorial Sloan-Kettering Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-050
Record Dates: First submitted 2005-08-17; First posted 2005-08-19 (Estimated); Last update posted 2008-12-23 (Estimated); Status verified 2008-12

CONDITIONS: Sarcoma
Keywords: IMRT+Surgery versus Surgery For Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Radiotherapy, Intensity-Modulated

INTERVENTIONS:
Procedure: Surgical Resection
Procedure: Intensity Modulated Radiation Therapy (IMRT)

SUMMARY:
This is a phase III clinical trial for patients with potentially completely resectable primary retroperitoneal sarcoma. Patients who take part will be divided into two groups, a radiation therapy plus surgery group and a surgery alone group.

Patients in the radiation therapy plus surgery group will receive radiation treatments as an outpatient. Surgery to try to remove the remaining tumor will be done after the radiation treatments are completed.

Patients in the surgery alone group will have surgery to try to remove all tumor.

DETAILED DESCRIPTION:
Primary Objective: To ascertain whether patients with completely resected (R0 + R1), primary retroperitoneal sarcoma who are randomized to pre-operative IMRT and surgery have a longer recurrence-free survival compared to patients randomized to treatment with surgery alone.

Secondary Objectives: To ascertain whether patients with completely resected (R0 + R1), primary retroperitoneal sarcoma randomized to pre-operative IMRT and surgery have longer overall survival compared to patients randomized to treatment with surgery alone.

* To compare the resectability rate between the two arms
* Determine the variability of NMR biochemical profiles and the variability of expression for genes/proteins involved in adipocyte differentiation, cell cycle control and apoptosis within different regions of the primary retroperitoneal sarcoma in patients treated with surgery alone and pre-operative radiotherapy.
* Analyze NMR biochemical patterns and expression patterns for genes/proteins involved in adipocyte differentiation, cell cycle control and apoptosis to identify markers that can provide an objective measure of sarcoma differentiation, proliferation, and apoptosis.
* Predict the response of sarcoma to radiation therapy and the risk of local recurrence, based on data derived from NMR biochemical and gene/protein expression patterns in patient tumors that recurred compared to those without recurrence.
* Determine if diffusion-weighted MRI early in course of radiation therapy can predict the ultimate pathologic response of sarcoma following resection and the risk of local recurrence.
* Analyze plasma levels of VEGF, FGF, Ang-1, Ang-2 and endostatin prior to and following therapy and correlate with treatment response, local and distant recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary retroperitoneal/pelvic soft tissue sarcoma.
* Gross total resection (RO or R1) must be feasible.
* No prior chemotherapy, immunotherapy or radiotherapy is allowable.
* Patients should be over 18 years of age and capable of providing informed consent indicating awareness of the investigational nature of this trial, in keeping with hospital policy.
* Karnofsky performance status of >= 70 %
* No other concurrent chemotherapy, immunotherapy or radiotherapy is allowable.
* Adequate organ function defined as follows: absolute granulocytes >= 1,500/mm 3, platelets >= 150,000/mm 3, serum bilirubin <= 1.5 mg/dl, serum creatinine <= 1.5 mg/dl.
* Written informed consent (study specific) must be obtained from each patient prior to entering the study.
* Patients should be willing to be followed at Memorial Sloan-Kettering Cancer Center during the course of treatment and follow-up.
* Patients must be able to get IMRT radiotherapy at Memorial Sloan-Kettering Cancer Center

Exclusion Criteria:

* Patients presenting with primary non-retroperitoneal soft tissue sarcoma or recurrent retroperitoneal sarcoma.
* Patients who are deemed unresectable by clinical/imaging criteria.
* Patients with histologic diagnosis of gastrointestinal stromal sarcoma, desmoplastic small round cell tumor, desmoid, Ewing's sarcoma, PNET, adenosarcoma, granular cell tumor, mesothelioma or rhabdomyosarcoma are excluded from the study.
* Patients with known metastatic disease, or those with radiologically evident metastases.
* Patients with clinically significant heart disease (NYHA Class III/IV), history of active angina or myocardial infarction within 6 months, history of significant ventricular arrhythmia requiring medication with antiarrhythmics or a history of clinically significant conduction system abnormality. Patients with any of the above conditions who are seen by a cardiologist at MSKCC and are found to be an acceptable risk for surgery will be allowed to participate in this study.
* Patients with any active concurrent malignancy other than non-melanoma skin cancers or carcinoma-in situ of the cervix. Patients with previous malignancies but without evidence of disease for > 5 years will be eligible.
* Women who are pregnant.
* Patients currently participating in other clinical trials the requirements of which may preclude their complete involvement in this study
* Patients with serious intercurrent infections or non-malignant uncontrolled illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2003-05; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
To ascertain whether patients with completely resected (R0 + R1), primary retroperitoneal sarcoma who are randomized to pre-operative IMRT and surgery have a longer recurrence-free survival compared to patients randomized to treatment with surgery alone.

SECONDARY OUTCOMES:
• To ascertain whether patients with completely resected (R0 + R1), primary retroperitoneal sarcoma randomized to pre-operative IMRT and surgery have longer overall survival compared to patients randomized to treatment with surgery alone.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Singer, M.D, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org